CLINICAL TRIAL: NCT06327789
Title: The Relationship Between Trunk Control and Disability in Persons With Early Relapsing Multiple Sclerosis
Brief Title: Trunk Control and Disability in Persons With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ARZUCAN TOKSAL, MSc physiotherapist, Zonguldak Bulent Ecevit University
Other Study IDs: ZBEU-MS
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: Patients who were 18-50 years old, diagnosed with RRMS by a experienced neurologist, and with an EDSS score ≤ 3 were included in this study. Patients with orthopedic or sensory additional problems in the lower extremity, who had an interventional procedure in the last six months, and had an attack in the last three months were excluded from the study.

SUMMARY:
This study aims to investigate the relationship between physical disability and trunk control, balance, and pedobarographic parameters in persons with Relapsing Remitting Multiple Sclerosis (RRMS) who have a low Expanded Disability Status Scale (EDSS) score. Twenty-three RRMS patients with an age range of 18-50 years, EDSS score ≤ 3 were included in this study. The patients' level of disability (EDSS), trunk control )Trunk Impairment Scale - TIS), lower extremity functionality (Timed 25-Foot Walk Test - T25FW), upper extremity functionality (Nine Hole Peg Test- 9HPT), balance (Biodex Balance System) and gait (Zebris® FDM 2) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old,
* diagnosed with RRMS by an experienced neurologist
* EDSS score ≤ 3

Exclusion Criteria:

* orthopedic or sensory additional problems in the lower extremity
* who had an interventional procedure in the last six months, and had an attack in the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: diagnosed with relapsing-remitting multiple sclerosis by an experienced neurologist
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | up to 8 weeks
  EDSS was used to determine the patients' level of disability. EDSS is most commonly used to assess the level of disability in persons with MS. In this scale pyramidal, cerebral, cerebellar, brainstem, visual and sensory subparameters are evaluated it consists of ordinal rating system ranging from 0 (normal neurological status) to 10 (death due to MS) in 0.5 increments interval (when reaching EDSS 1). The lower scale values of the EDSS measure impairments based on the neurological examination, while the upper range of the scale (> EDSS 6) measures handicaps of patients with MS. The determination of EDSS 4 - 6 is heavily dependent on aspects of walking ability
Trunk Impairment Scale (TIS) | up to 8 weeks
  This scale used to evaluate the trunk control of the participants, TIS contains static sitting balance, dynamic sitting balance, and coordination. The total score of this scale is from 0 to 23 and a high score indicates better trunk control. The patients were placed in the standard sitting position for the test and the parameters were applied. Standart position is such that the knees are flexed at 90 degrees, without back support, with the hands and forearms on the thighs and the feet in contact with the ground.
Biodex Balance System (BBS) (MedicalSystems, Shirley, NY, USA) | up to 8 weeks
  This system is a multiaxial device that objectively measures and records a patient's ability to stabilize the involved joint under dynamic stress. The BBS measures, in degrees, the tilt about each axis during dynamic conditions and calculates a medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and an overall stability index (OSI). These indexes represent fluctuations around a zero point established before testing when the platform is stable. A high score in the all parameters indicates poor balance. The test was performed in 3 repetitions, each lasting 20 seconds, with a 10-second rest period in between, under different conditions, including eyes open-closed, firm-foam surface, and static-dynamic surface. The average of the three repetitions was calculated automatically by the device
Step Length (cm) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Stride Length (cm) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Step Width (cm) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Cadence (steps/min) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Velocity (m/s) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Step time (s) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Stride time (s) | up to 8 weeks
  The temporal-spatial characteristics of gait were assessed through the utilization of dynamic pedobarography. Dynamic pedobarographic analysis was performed with the implementation of a pressure platform (Zebris® FDM 2, dimensions 212.2x60.5x2.5 cm, Zebris Medical GmbH, Germany) positioned at the center of an 8-meter walking path. Patients completed the gait cycle three times, once for forward and once for backward gait, while barefoot.
Timed 25-Foot Walk Test (T25FW) | up to 8 weeks
  This test is designed for the evaluation of lower extremity functions.Initiated at the participant's first step, the test concludes upon reaching the finish line. The participants are instructed to walk as expeditiously as feasible within a specified time frame without running. The duration taken to traverse the 25-foot distance, both for the outbound and return segments, is documented, and subsequently, the average of these two durations is calculated.
Nine-Hole Peg Test (9HPT) | up to 8 weeks
  It is a short, standardized, quantitative test used to evaluate upper extremity function. In the test, patients are asked to pick up nine wooden pegs from a platform as quickly as possible and then place them back into the holes.In our study, the test was conducted twice for both the dominant and non-dominant hands, and the average completion time was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Piri Çınar, Principal Investigator — Samsun University; Güngör Beyza Özvar Şenöz, Principal Investigator — Yüksek İhtisas University; Hasret Uçar, Principal Investigator — Zonguldak Bulent Ecevit University; Serkan Özakbaş, Principal Investigator — Dokuz Eylul University; Mustafa Açıkgöz, Principal Investigator — Zonguldak Bulent Ecevit University; Nursena Ceylan, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)